CLINICAL TRIAL: NCT00972114
Title: Coronary Artery Bypass Graft Surgery Combined Pedicled Omentum Wrapped Autologous Atrial Tissue Patch Cardiomyoplasty for Patients With Ischemic Cardiomyopathy: a Prospective Randomized Controlled Clinical Trial
Brief Title: CABG Combined Pedicled Omentum Wrapped Autologous Atrial Tissue Patch Cardiomyoplasty for Ischemic Cardiomyopathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Shengshou Hu MD, FACC, China National Center for Cardiovascular Diseases
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20090903
Record Dates: First submitted 2009-09-03; First posted 2009-09-04 (Estimated); Last update posted 2009-12-10 (Estimated); Status verified 2009-12

CONDITIONS: Ischemic Cardiomyopathy; Congestive Heart Failure; Coronary Artery Disease
MeSH Terms: conditions — Heart Failure; Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CABG combined cardiomyoplasty (Experimental): Coronary artery bypass graft surgery combined pedicled omentum wrapped autologous atrial tissue patch cardiomyoplasty
  Interventions: Procedure: CABG combined cardiomyoplasty
- CABG combined pedicled omentum graft (Active Comparator): Coronary artery bypass graft surgery combined pedicled omentum graft
  Interventions: Procedure: CABG combined pedicled omentum graft
- CABG alone (Active Comparator): Coronary artery bypass graft surgery alone
  Interventions: Procedure: CABG alone

INTERVENTIONS:
Procedure: CABG combined cardiomyoplasty — coronary artery bypass graft surgery combined pedicled omentum wrapped autologous atrial tissue patch cardiomyoplasty
  Other Names: CABG combined pedicled omentum graft
  Arms: CABG combined cardiomyoplasty
Procedure: CABG combined pedicled omentum graft — Coronary artery bypass graft surgery combined pedicled omentum graft
  Arms: CABG combined pedicled omentum graft
Procedure: CABG alone — Coronary artery bypass graft surgery alone
  Other Names: Coronary artery bypass graft surgery alone
  Arms: CABG alone

SUMMARY:
The purpose of this study is in a phase I/II safety and efficacy study to evaluate the clinical effect of coronary artery bypass graft (CABG) combined pedicled omentum wrapped autologous atrial tissue patch cardiomyoplasty for patients with ischemic cardiomyopathy.

DETAILED DESCRIPTION:
This is a phase I/II, randomized controlled trial to evaluate the use of CABG combined pedicled omentum wrapped autologous atrial tissue patch cardiomyoplasty for patients with ischemic cardiomyopathy. The study hypothesis is that the combined surgical technique to perform pedicled omentum wrapped autologous atrial tissue patch cardiomyoplasty as adjunct to CABG, is safe to patients with severe ischemic heart failure and can improve regional myocardial perfusion contractility, which resulting in improved systolic and diastolic left ventricular function.

The primary object of this study will be to evaluate the safety and efficacy of this novel combined surgical technique. The efficacy will be assessed changes in left ventricular ejection fraction by MRI. The secondary endpoint of the study is to assess the effects of this novel combined surgical technique on cardiac contractile function and functional outcome. The effects will be assessed on the basis of clinical status and imaging rests in 6 month follow-up after enrollment. A maximum of 60 patients between 20 and 70 years will be enrolled in the study. These participants will be randomized to receive CABG, pedicled omentum graft combined CABG, or pedicled omentum graft autologous atrial tissue patch cardiomyoplasty combined CABG. The objective evaluations will be performed at baseline and during 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* 20-70 years old;
* Ability to give informed consent;
* Documented severe coronary heart disease, defined as at least 70% luminal diameter narrowing of at least three major coronary artery, suited to CABG;
* Left ventricular dysfunction (LVEF) less than or equal to 35%, measured by MRI or less than or equal to 45%, measured by echocardiogram;
* Presence of reversibility, as identified by single photon emission computed tomography (SPECT) isotope protocol;
* At least 3 months since last episode of myocardial infarction;
* Without a history of abdominal operation and severe abdominal diseases;
* Negative pregnancy test (in women with childbearing potential.

Exclusion Criteria:

* Pregnant or lactating;
* A history of malignancy in the last 5 years excluding basal cell carcinoma, that has been surgically removed, with proof of surgical clean margins;
* a history of abdominal operation or severe abdominal diseases;
* Positive test result for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
* Any condition requiring immunosuppressive medication;
* Bleeding diathesis, defined as an international normalized ratio of at least 2.0 in the absence of warfarin therapy;
* Hepatic dysfunction, as defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 1.5 times the upper limit of normal range prior to study entry;
* Chronic renal insufficiency, defined as a serum creatinine level greater than 2.5 mg/dL or requiring dialysis;
* Leukocytes less than 4,000/µL or exceeding 10,000/µL;
* Platelets less than 100,000/µL;
* Hemoglobin less than 10 g/dL;
* Chronic atrial fibrillation;
* Less than 3 months since last episode of cerebral infarction;
* Implantable cardioverter-defibrillator shock within 30 days of baseline consent, and within 30 days of randomization;
* Presence of ventricular tachycardia lasting 30 seconds or more on 24-hour Holter monitor or electrocardiogram (ECG) performed during screening period;
* Patients for whom it is impossible to perform both cardiac MRI;
* Enrolled in an investigational device or drug study within the previous1 year;
* Any other reason that the Clinical Supervisors or Clinical Researchers may have for considering a case unsuitable for the study.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-06 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Safety of CABG combined pedicled omentum wrapped autologous atrial tissue transplantation. | 6 months
Changes in left ventricular ejection fraction (LVEF) by MRI. | 6 months

SECONDARY OUTCOMES:
Changes in LVEF by echocardiography. | 6 months
Changes in regional wall motion by MRI. | 6 months
Changes in regional wall motion by echocardiography. | 6 months
Changes in fixed perfusion defect(s) by single photon emission computed tomography. | 6 months
Clinical improvements, including change in 6 minutes walk test, as determined by multiple measures. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shengshou Hu, MD, Study Director — National Center for Cardiovascular Diseases, China
Locations (2):
- China (2):
  - China National Center for Cardiovascular Diseases, Cardiovascular Institute & Fuwai Hospital, Beijing
  - Institute of cardiovascular diseases & Fuwai hospital, Beijing